CLINICAL TRIAL: NCT06898658
Title: Mindfulness and Cardiometabolic Health for Spanish Speaking Latina Pregnant Women: A Community-informed Project Targeting Inflammatory Gene Expression and Glycemic Control
Brief Title: Conscious Pregnancy: Supporting Maternal Cardiometabolic Health With Mindfulness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lauren Gyllenhammer, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4967; P50MD017344 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-03-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Maternal Cardiometabolic Health; Molecular Impact of Psychological Stress and Socioeconomic Adversity; Maternal Inflammatory Markers; Maternal Diabetes; Maternal Behavior; Maternal Distress
MeSH Terms: conditions — Financial Stress; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait-List Control Group (No Intervention): Participants randomized to control will continue their usual care (MOMS at-home visitation schedule) and will provide concordant pre- and post-intervention data alongside the intervention group. They will receive audio recordings of all mindfulness instructional material after the 6-week intervention and post-intervention data collection is complete.
- Mindfulness Intervention Group (Experimental): The culturally tailored mindfulness program will be delivered in a hybrid format and is an adaptation of the validated Mindfulness Awareness Practices (MAPs), which has been utilized in Spanish speaking Latino populations and in the context of pregnancy. MAPs trains one in the systematic practice of attending to moment-by-moment experiences, thoughts, and emotions from a nonjudgmental perspective, and is more accessible to diverse and socioeconomically disadvantaged populations relative to standard mindfulness-based Interventions, as it does not require a day-long retreat or yoga practice.
  Interventions: Behavioral: Mindfulness Intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Hybrid MAPs course will be delivered by a Spanish-speaking Latina certified mindfulness instructor, with a blend of in-person instruction, online instruction and asynchronous (audio-recorded) content instruction over 6-wks. There will be three live-2hr classes (2 in-person, 1 online) and three 3 weeks of 1-hr self-guided audio/week asynchronous content (1hr/wk). Additionally, the instructor will invite the intervention group to join optional weekly via Zoom 1x/wk for 30-min sessions for time to encourage questions, dialogue, and brief group mindfulness practice opportunities.
  Class attendance and engagement with audio-recorded materials will be tracked. The study team will call or text participants weekly to maintain engagement, remind about any upcoming scheduled classes, and answer any questions. Participant attendance in classes (in-person and zoom) will be monitored.
  Arms: Mindfulness Intervention Group

SUMMARY:
A pilot randomized control trial (RCT) to examine the efficacy of a culturally tailored mindfulness intervention upon fasting cardiometabolic factors (including markers of glycemic control) and inflammatory gene expression in n=60 (n=30 intervention, n=30 wait-list control) low-income Spanish-speaking Latina pregnant women. The study will be conducted in partnership with MOMS, a nonprofit community organization that serves low-income pregnant and postpartum women.

DETAILED DESCRIPTION:
Prenatal health interventions have the potential to shape the future health of both mothers and offspring. Given that the Latino population is disproportionately affected by high rates of obesity and type 2 diabetes, targeted prenatal health interventions that support Latina metabolic health are fundamental to reduce the burden of Latino health disparities within and across generations. Research in primarily non-Hispanic White populations suggests that prenatal mindfulness interventions can not only improve maternal mental health outcomes and well-being, but additionally can support systemic physiological health, such as improved glycemic control and reduced gestational weight gain. However, research on the acceptability and feasibility of mindfulness programs for Latino populations is limited, especially among those who are Spanish-speaking and affected by poverty. Focus groups conducted with this target population, have highlighted a strong interest in mindfulness programs, with a need for novel hybrid instruction format (live classes + digital at-home content). Accordingly, the investigators have developed an adapted, hybrid version of the validated 6-week Mindfulness Awareness Practices (MAPs) training program in Spanish and English.

Here, the investigators plan to pilot and examine the efficacy of this culturally tailored mindfulness intervention upon cardiometabolic factors, including inflammatory gene expression and glycemic control markers, in a low-income Spanish-speaking Latina pregnant population (n=60; n=30 intervention, n=30 wait-list control). Specifically, the investigators will examine the intervention impact on cardiometabolic markers (e.g., fasting glucose and insulin, Hemoglobin A1c (HbA1c), C-reactive protein (CRP), lipids), and inflammatory gene expression measurement. Maternal mental well-being, pregnancy and birth outcomes will also be assessed. In addition, the investigators will examine the feasibility and acceptability of pre-post intervention continuous glucose monitoring (CGM) in n=5 mindfulness group participants.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton, intrauterine pregnancy
2. 1st or 2nd trimester at enrollment
3. Fluent in Spanish
4. Self-identify as Hispanic/Latino
5. Low-income

Exclusion Criteria:

1. Having regular mindfulness practice
2. T1 or T2D diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maternal Pro-Inflammatory Gene Expression | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  The primary outcome is maternal pro-inflammatory gene expression, as determined from pre-post intervention change in pre-specified transcriptional regulation factors from the conserved transcriptional response to adversity (CTRA) (e.g., proinflammatory nuclear factor κB (NF-κB)). Gene expression will be quantified from dried blood spots (DBS). Comparison of intervention and control group will occur pre and post mindfulness intervention.
High Sensitivity C-Reactive Protein | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  High sensitivity c-reactive protein (hs-CRP) is a circulating marker of systemic inflammation. hs-CRP will be measured in dried blood spots (DBS) and reported in mg/L units.
Fasting Glucose | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Fasting glucose will be measured using a glucometer and reported in mg/dL.
Hemoglobin A1c (HbA1c) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Hemoglobin A1c (HbA1c) will be measured in DBS and reported as a percentage (%), which indicates the proportion of hemoglobin molecules that are coated with glucose.
Fasting Insulin | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Fasting insulin will be measured via DBS and reported in uIU/mL units.
Lipid Panel | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Fasting apolipoprotein A (ApoA1), apolipoprotein B (ApoB), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), total cholesterol, and triglycerides will be collected via DBS and reported in mg/dL units.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Perceived stress will be measured using the validated 4-item perceived stress scale (PSS), with a higher score indicated greater perceived stress (scale range 0-16).
Edinburgh Postnatal Depression Scale (EPDS) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Depressive symptomatology will be measured with the validated 10-item Edinburgh Postnatal Depression Scale (EPDS). A higher score indicates greater depressive symptomatology and a score >= 13 indicates high risk for depression (scale range 0-30).
Five Facet Mindfulness Questionnaire (FFMQ) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  The validated15-item five facet mindfulness questionnaire (FFMQ) will be used to assess mindfulness, with a higher score indicating greater mindfulness with regards to thoughts, experiences, and actions in daily life (scale range 15-75).
Pregnancy-related anxiety (PRAQ-R2) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  The validated 10-item pregnancy-related anxiety scale revised-2 (PRAQ-R2) will be used to assess prenatal anxiety, with higher scores indicating greater pregnancy-related anxiety (scale range 10-50).
State-Trait Anxiety Inventory (STAI) | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  State anxiety will be measured using the validated state-trait anxiety inventory (STAI). The state anxiety subscale will quantify the perceptions of anxiety in the present moment, with higher scores indicating greater self-report of anxiety (scale range 6-24).
Spot Morning Cortisol Sample | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Fasting morning cortisol will be measured in DBS and reported in ug/dL units. Time since waking will be recorded and accounted for in analyses.
Homocysteine | Comparison of intervention and control group will occur pre and post 6-week mindfulness intervention
  Homocysteine will be measured via DBS and reported in umol/L units. Higher homocysteine levels are linked to increased inflammation.

OTHER OUTCOMES:
Acceptability of Continuous Glucose Monitoring (CGM) | 8 weeks (1 week of measurement prior to starting 6 week intervention, and 1 week measurement after intervention completion))
  Masked upper arm continuous glucose monitoring (CGM) monitoring 1-week pre-post intervention will be assessed in a subsample (n=5 mindfulness group), using Dexcom G6. Acceptability of the 1-week GCM data will be determined by the post collection survey report of acceptability and number of adverse event reporting (e.g., skin irritation).
Feasibility of CGM | 8 weeks (1 week of measurement prior to starting 6 week intervention, and 1 week measurement after intervention completion))
  Feasibility of the 1-week GCM data will be determined by the enrollment rate (enrollment offered on a rolling basis to all mindfulness participants, enrollment rate will be calculated as number of invitations required to achieve consent in n=5), and number of days with complete data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Gyllenhammer, PhD, Principal Investigator — University of California, Irvine; Karen L Lindsay, RD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- MOMS, Santa Ana, California, United States

IPD SHARING:
Plan to Share IPD: No